CLINICAL TRIAL: NCT05011994
Title: Maintenance of Physical Activity After Cardiac Rehabilitation: a Feasibility Trial
Brief Title: Maintenance of Physical Activity After Cardiac Rehabilitation
Acronym: FAIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Slagelse Hospital (Other)
Collaborators: City of Slagelse (municipality) (Unknown); Holbaek Sygehus (Other); University of Southern Denmark (Other); University College Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EMN-2021-00020; EMN-2021-00020 (Other: Research Ethics Committee of Region Zealand, Denmark); REG-162-2020 (Other: Danish Data Protection Agency through Region Zealand)
Record Dates: First submitted 2021-07-17; First posted 2021-08-19 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Ischemia; Heart Failure; Arrythmia; Heart Arrest
Keywords: cardiac rehabilitation; ischemic heart disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Myocardial Ischemia; Heart Failure; Arrhythmias, Cardiac; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maintenance intervention (Experimental): Participants will receive a 12-week mobile health (mHealth) intervention that consists of action planning, text messages, and coordinator support.
  Interventions: Behavioral: Maintenance intervention

INTERVENTIONS:
Behavioral: Maintenance intervention — The intervention consists of action planning, text messages, and coordinator support.
  At onset, each participant creates an action plan for physical activity with the help of a health professional:
  * What types of physical activities?
  * When and how often?
  * Where and with who?
    2 auto-generated text messages are sent weekly for a duration of 12 weeks. The first prompts physical activity. The second asks if plans were reached. If yes, an automatic reply with positive reinforcement is generated. If no, an automatic reply asks if the participant wants to be contacted.
  Participants are contacted by a coordinator either by answering text messages or if not answering the texts for a period of 2 weeks or more. Coordinator functions:
  * Call participants replying to texts that they wish to be contacted
  * Help participants establish contact to local activities involving physical activity
  * Follow-up on and adjustment of action plan
  * Offer guidance in physical activity

SUMMARY:
Physical activity is a key element in cardiac rehabilitation and prevention of cardiovascular mortality and hospitalizations. After cardiac rehabilitation programs end, physical activity levels and participation in continued cardiac rehabilitation declines. The aim of this study is to evaluate the feasibility a mobile health intervention with text messages and behavior change theory in patients with cardiovascular disease for a duration of 3 months after completion of a cardiac rehabilitation program. An intervention consisting of action planning, text messages, and coordinator support is tested in a feasibility trial design with 40 expected participants.

DETAILED DESCRIPTION:
Physical activity is a key element in cardiac rehabilitation and prevention of cardiovascular mortality and hospitalizations. After cardiac rehabilitation programs end, physical activity levels and participation in continued cardiac rehabilitation declines.

The primary aim of this study is to evaluate the feasibility in terms of recruitment, retention, data completeness, intervention delivery and compliance, and acceptability of a mobile health intervention with text messages and behavior change theory in patients with cardiovascular disease for a duration of 3 months after completion of a cardiac rehabilitation program.

The study is a single-group multi-site feasibility trial. Participants will be recruited from phase II cardiac rehabilitation programs at Slagelse Hospital, the city of Slagelse (municipality), and Holbæk Hospital. Starting immediately after completion of cardiac rehabilitation, study participants will receive an intervention that consists of action planning, text messages, and coordinator support for a period of 12 weeks (see more details under 'Arms and Interventions'). The investigators base the intervention on a theoretical model of behavior change in the form of the Health Action Process Approach (HAPA). Behavior change techniques (BCTs) are used as part of the intervention. The intervention is an addition to standard practice and does not replace any existing treatment offers.

To evaluate the feasibility of the intervention and its readiness to be tested in a subsequent RCT design, the investigators have set progression criteria using a system of green (proceed to RCT), amber (amend when proceeding to RCT), or red (issue must be solved before proceeding to RCT). The progression criteria are listed under 'Primary Outcome Measures'.

Participants will wear accelerometers on thigh and wrist for 1 and 3 weeks, respectively, starting 1 week before end of cardiac rehabilitation. Baseline measurements and start of intervention is planned to be at the same time as cardiac rehabilitation ends. After 11 weeks of intervention, participants will attend a follow-up assessment, where participants will wear accelerometers on thigh and wrist again.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Participant in an exercise-based cardiac rehabilitation program in either hospital or municipality setting.
* Access to a personal mobile phone and Danish telephone number.
* Able to walk 3 meters without assistance.

Exclusion Criteria:

* Insufficient Danish language proficiency to read and understand text messages and questionnaires.
* Patients cognitively or mentally unable to participate.
* Terminal patients and patients with a life expectancy of less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Baseline
  Green: Mean of ≥0.75 recruited participants per week per site
  Amber: Mean of 0.5-0.74 recruited participants per week per site
  Red: Mean of <0.5 recruited participants per week per site
Attrition/retention through follow-up assessment session | Up to 12 weeks
  Green: ≥80% retention of participants through follow up
  Amber: 50-79% retention of participants through follow up
  Red: <50% retention of participants through follow up
Accelerometer data completeness | Baseline
  Green: Accelerometer data from both baseline and follow-up available on ≥80% of completing participants
  Amber: Data available on 50-79% of completing participants
  Red: Data available on <50% of completing participants
Accelerometer data completeness | 12 weeks
  Green: Accelerometer data from both baseline and follow-up available on ≥80% of completing participants
  Amber: Data available on 50-79% of completing participants
  Red: Data available on <50% of completing participants
Response rate on patient reported outcomes | Baseline
  Green: ≥90% of participants attending baseline and follow-up assessment return patient reported outcomes
  Amber: 75-89% of patients attending baseline and follow-up assessment return patient reported outcomes
  Red: <75% of participants attending baseline and follow-up assessment return patient reported outcomes
Response rate on patient reported outcomes | 12 weeks
  Green: ≥90% of participants attending baseline and follow-up assessment return patient reported outcomes
  Amber: 75-89% of patients attending baseline and follow-up assessment return patient reported outcomes
  Red: <75% of participants attending baseline and follow-up assessment return patient reported outcomes
Coordinator time spent, minutes per participant throughout the intervention | 12 weeks
  Green: Mean coordinator time spent of ≤30 minutes per participant
  Amber: Mean coordinator time spent of 31-60 minutes per participant
  Red: Mean coordinator time spent of >60 minutes per participant
Response rate (adherence) to weekly follow-up messages | 12 weeks
  Green: ≥75% of patients respond to at least 75% of messages
  Amber: 50-74% of patients respond to at least 75% of messages
  Red: <50% of patients respond to at least 75% of messages
Acceptability of text message component, single item | 12 weeks
  Green: ≥75% of participants find text messages acceptable
  Amber: 50-74% of participants find text messages acceptable
  Red: <50% of participants find text messages acceptable

SECONDARY OUTCOMES:
Physical activity, objectively measured | Change from baseline to 12 weeks
  Measured with thigh and wrist accelerometers
Physical function, walking | Change from baseline to 12 weeks
  6 minute walking test
Physical function, sit-to-stand | Change from baseline to 12 weeks
  30-second sit-to-stand test
Physical activity, subjectively measured | Change from baseline to 12 weeks
  The International Physical Activity Questionnaire (IPAQ) is used to measure physical activity in the past 7 days. 0 is minimum (completely inactivty).

OTHER OUTCOMES:
Health-related quality of life, general | Change from baseline to 12 weeks
  EQ-5D-5L evaluates health status in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated from 1 (best) to 5 (worst) and overall health is rated on a 0 to 100 VAS scale.
Health-related quality of life, VAS subscale | Change from baseline to 12 weeks
  EQ-5D-5L evaluates health status in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated from 1 (best) to 5 (worst) and overall health is rated on a 0 to 100 VAS scale.
Health-related quality of life, heart-specific | Change from baseline to 12 weeks
  HeartQoL is used to measure heart-specific quality of life in the past 4 weeks. Range from 0 (worst) to 42 (best) .
Anxiety and depression | Change from baseline to 12 weeks
  Hospital Anxiety and Depression Scale (HADS). HADS gives a score for each of anxiety and depression, each ranging from 0 (best) to 21 (worst).
Physical function, self-reported | Change from baseline to 12 weeks
  WHO Disability Assessment Schedule 2.0 (WHODAS 2.0),12-item version. WHODAS is a generic assessment instrument for health and disability. Range from 12 (no disability) to 60 (highest disability or loss of function).
Comorbidity | Change from baseline to 12 weeks
  Disease Burden: Morbidity Assessment by Self-Report used to evaluated a list of common chronic conditions affect the participants' daily activities. Each condition (that the participant has) is rated from 1 (not at all) to 5 (a lot) in regard to how much it limits daily activities.
Self-efficacy, managing chronic disease | Change from baseline to 12 weeks
  Self-efficacy of managing chronic disease 6 items scale. Score is calculated as the mean of 6 items, each scored from 1 (low self-efficacy) to 10 (high self-efficacy).
Motivational Self-efficacy | Change from baseline to 12 weeks
  Motivational self-efficacy, HAPA items by Schwartzer R., 2 items each rated on a scale from 1 (low self-efficacy) to 4 (high self-efficacy).
Coping Self-efficacy | Change from baseline to 12 weeks
  Coping self-efficacy, HAPA items by Schwartzer R., 2 items each rated on a scale from 1 (low self-efficacy) to 4 (high self-efficacy).
Recovery Self-efficacy | Change from baseline to 12 weeks
  Recovery self-efficacy, HAPA items by Schwartzer R., 2 items each rated on a scale from 1 (low self-efficacy) to 4 (high self-efficacy).

CONTACTS AND LOCATIONS:
Overall Officials: Rune M Andersen, PhD, Principal Investigator — Næstved-Slagelse-Ringsted Hospitals; University of Southern Denmark; Lars H Tang, PhD, Study Chair — Næstved-Slagelse-Ringsted Hospitals; University of Southern Denmark; Søren T Skou, PhD, Study Chair — Næstved-Slagelse-Ringsted Hospitals; University of Southern Denmark
Locations (3):
- Denmark (3):
  - Holbæk Hospital, Holbæk
  - City of Slagelse (municipality), Korsør
  - Slagelse Hospital, Slagelse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen RM, Skou ST, Clausen MB, Jager M, Zangger G, Grontved A, Brond JC, Soja AMB, Tang LH. Maintenance of physical activity after cardiac rehabilitation (FAIR): study protocol for a feasibility trial. BMJ Open. 2022 Apr 5;12(4):e060157. doi: 10.1136/bmjopen-2021-060157. PMID 35383088
- See also: Link to published study protocol — https://bmjopen.bmj.com/content/12/4/e060157.info